CLINICAL TRIAL: NCT07197008
Title: Sacituzumab Tirumotecan (Sac-TMT) Plus Bevacizumab in 3rd Generation EGFR-TKI Treated Advanced EGFR-mutant Nonsquamous NSCLC With Brain Metastasis: a Single-arm, Phase II Study（TOP BRAIN）
Brief Title: Sacituzumab Tirumotecan (Sac-TMT) Plus Bevacizumab in 3rd Generation EGFR-TKI Treated Advanced EGFR-mutant Nonsquamous NSCLC With Brain Metastasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li-kun Chen (Other)
Responsible Party: Sponsor-Investigator, Li-kun Chen, doctor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-287
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: brain metastases; EGFR mutated; Sacituzumab tirumotecan
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible patients will receive SKB264 at a dose of 4 mg/kg in combination with bevacizumab 5mg/kg by intravenous infusion on day 1 and day 15 of each 28-day cycle. All enrolled participants will continue to receive the study treatment until disease progression or unacceptable toxicity or patient requests to discontinue the treatment, whichever occurs first.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab tirumotecan plus bevacizumab (Experimental): Eligible patients will receive Sacituzumab tirumotecan at a dose of 4 mg/kg in combination with bevacizumab 5mg/kg by intravenous infusion on day 1 and day 15 of each 28-day cycle. All enrolled participants will continue to receive the study treatment until disease progression or unacceptable toxicity or patient requests to discontinue the treatment, whichever occurs first. Tumor evaluation for intracranial and extracranial lesions was independently assessed by investigators. Imaging assessments will be conducted every 6 weeks (±1 week) for the first 48 weeks, and thereafter every 8 weeks (±1 week) until disease progression, initiation of a new antitumor treatment, withdrawal of consent, loss to follow-up, death, or the end of the study, whichever occurs first.
  Interventions: Drug: Sacituzumab tirumotecan (Sac-TMT) plus bevacizumab

INTERVENTIONS:
Drug: Sacituzumab tirumotecan (Sac-TMT) plus bevacizumab — Eligible patients will receive Sacituzumab tirumotecan at a dose of 4 mg/kg in combination with bevacizumab 5mg/kg by intravenous infusion on day 1 and day 15 of each 28-day cycle.

SUMMARY:
This is a prospective, single-center, phase 2 clinical study to explore the efficacy and safety of Sac-TMT in combination with bevacizumab for patients with EGFR-mutated nonsquamous NSCLC with brain metastases. The study will enroll 50 EGFR-sensitive mutation(19del/21L858R) nonsquamous NSCLC patients who progressed on or after 3rd generation EGFR-TKI with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤80 when signing the informed consent form, regardless of gender;
2. Histologically or cytologically confirmed nonsquamous NSCLC with EGFR-sensitive mutation (exon 19 deletion or exon 21 L858R mutation).
3. Progression on or after 3rd-generation EGFR-TKI (change to the third-generation EGFR-TKIs after receiving 1st or 2nd generations of TKI, or to use the third-generation TKI in the first line are all allowed).
4. Brain parenchymal metastases confirmed by cranial MRI, including asymptomatic BM or those with symptoms controlled after local treatment and/or dehydration therapy, should maintain a clinically stable state (no longer requiring glucocorticoids or anticonvulsants) for at least 2 weeks before the first dose.
5. According to mRECIST 1.1, the subject must have at least one accurately measurable intracranial target lesion that has not been previously treated with local therapies such as radiation therapy or surgery. Brain metastatic lesions with a diameter of ≥ 5 mm are permitted to be designated as target lesions.
6. ECOG PS 0-1.
7. Estimated life expectancy of 12 weeks or more.
8. Adequate organ function.
9. Female subjects of childbearing potential and male subjects whose partners are of childbearing potential must agree to use effective medical contraceptive measures from the time of signing the informed consent form until 6 months after the last dose.
10. The subject voluntarily participates in this study, signs the informed consent form, and is able to comply with the study visits and related procedures as specified in the protocol.

Exclusion Criteria:

1. Histologically or cytologically confirmed tumor with components of small cell lung cancer, neuroendocrine carcinoma, carcinosarcoma, or squamous cell carcinoma;
2. Patients with spinal cord compression or those assessed by the investigator as having extensive meningeal metastasis;
3. Previous whole-brain radiotherapy for brain metastases;
4. Subjects who have previously received chemotherapy, TROP2-targeted therapy, or any drug therapy containing topoisomerase I inhibitors, including antibody-drug conjugate (ADC) therapy (including in the context of adjuvant or neoadjuvant therapy);
5. Tumor invading or surrounding important surrounding organs and blood vessels (such as the heart, esophagus, superior vena cava, etc.), or with obvious necrosis, cavitation, or at risk of developing esophagotracheal fistula or esophagopleural fistula;
6. A history of bleeding tendency or coagulation disorder and/or clinically significant bleeding symptoms or risks within 4 weeks before the first dose;
7. Use of aspirin (> 325 mg/day) or treatment with dipyridamole or clopidogrel within 2 weeks before the first dose;
8. Use of full-dose oral or intravenous anticoagulants or thrombolytics within 2 weeks before the first dose;
9. Biopsy or other minor surgeries (excluding placement of vascular access devices) within 7 days before the first dose;
10. Presence of non-healing wounds or untreated fractures (excluding old fractures and other fractures that do not require treatment);
11. History of other malignant tumors within 3 years before the first dose (except tumors cured by local treatment, such as cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in situ, etc.);
12. Presence of any of the following cardiovascular and cerebrovascular diseases or risk factors:

    1. Myocardial infarction, unstable angina pectoris, acute or persistent myocardial ischemia, grade 3 or 4 heart failure (according to the New York Heart Association (NYHA) classification), symptomatic or poorly controlled severe arrhythmia, cerebrovascular accident, transient ischemic attack, or other severe cardiovascular and cerebrovascular diseases within 6 months before the first dose;
    2. Previous history of myocardial diseases such as myocarditis, primary cardiomyopathy, or specific cardiomyopathy;
    3. Any deep vein thrombosis within 3 months before the first dose (subjects with stable condition after treatment with low-molecular-weight heparin or drugs with similar effects for ≥ 2 weeks are permitted to enroll), peripheral arterial thromboembolic events, pulmonary embolism, or other severe thromboembolic events;
    4. Presence of major vascular diseases that may be life-threatening or require surgery within 6 months before the first dose, such as aortic aneurysm or aortic dissecting aneurysm;
13. Uncontrolled systemic diseases as judged by the investigator:
14. History of (non-infectious) interstitial lung disease (ILD) or non-infectious pneumonia requiring steroid treatment, current ILD or non-infectious pneumonia, or suspected ILD or non-infectious pneumonia at screening that cannot be excluded by imaging examinations;
15. Documented history of severe dry eye syndrome, severe meibomian gland disease and/or blepharitis, or severe corneal diseases that may impede/delay corneal healing;
16. Clinically severe lung damage caused by concurrent pulmonary diseases, including but not limited to any underlying lung diseases (such as severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease within 3 months before the first dose) or any autoimmune, connective tissue, or inflammatory diseases that may involve the lungs (i.e., rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc.), or previous pneumonectomy;
17. Subjects with active chronic inflammatory bowel disease, gastrointestinal obstruction, severe ulcer, gastrointestinal perforation, abdominal abscess, or acute gastrointestinal bleeding;
18. Proteinuria, evidenced by protein > 1.0 gram in urine test strip or 24-hour urine collection. All patients with protein ≥ 2+ in baseline urine test strip analysis must undergo 24-hour urine collection, and the protein in 24 hours must be proven to be ≤ 1 g;
19. Toxicity from previous anti-tumor treatment has not recovered to ≤ grade 1 (assessed based on NCI CTCAE v5.0) or the level specified in the inclusion/exclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
intracranial objective response rate | 6-months
  proportion of patients with complete or partial response of intracranial lesions

SECONDARY OUTCOMES:
intracranial progression-free survival | 12-months
  time from enrollment to intracranial disease progression or death.
systemic objective response rate | 6-months
  proportion of patients with complete or partial response of overall lesions
progression-free survival | 12-months
  time from enrollment to systemic disease progression [intracranial or extracranial or both] or death
overall survival | 36-months
  time from enrollment to death from any cause
adverse events | 12-months
  the incidence rate of adverse events according to CTCAE 5.0

IPD SHARING:
Plan to Share IPD: No